CLINICAL TRIAL: NCT00070564
Title: Phase III Trial of Continuous Schedule AC + G vs. Q 2 Week Schedule AC, Followed by Paclitaxel Given Either Every 2 Weeks or Weekly for 12 Weeks as Post-Operative Adjuvant Therapy in Node-Positive or High-Risk Node-Negative Breast Cancer
Brief Title: S0221 Adjuvant Doxorubicin, Cyclophosphamide, and Paclitaxel in Treating Patients With Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000334899; S0221 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IA breast cancer; stage IB breast cancer; stage IIIC breast cancer; male breast cancer; HER2-positive breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — pegfilgrastim; Cyclophosphamide; Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm I (Active Comparator): (closed 11/10/10) Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim subcutaneously (SC) on day 2 or filgrastim (G-CSF) SC on days 3-10. Treatment repeats every 14 days for 6 courses. Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 3 hours on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.
  Interventions: Biological: pegfilgrastim; Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Arm II (Experimental): (closed 11/10/10) Patients receive doxorubicin IV on day 1, oral cyclophosphamide on days 1-7, and G-CSF SC on days 2-7. Treatment repeats every 7 days for 15 courses. Beginning 2 weeks after completion of cyclophosphamide, patients receive paclitaxel and pegfilgrastim as in arm I.
  Interventions: Biological: pegfilgrastim; Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Arm III (Active Comparator): (closed 11/10/10) Patients receive doxorubicin, cyclophosphamide, and pegfilgrastim or G-CSF as in arm I. Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 1 hour on day 1. Treatment repeats every 7 days for 12 courses.
  Interventions: Biological: pegfilgrastim; Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Arm IV (Experimental): (closed 11/10/10) Patients receive doxorubicin, cyclophosphamide, and G-CSF as in arm II. Beginning 2 weeks after completion of cyclophosphamide, patients receive paclitaxel as in arm III.
  Interventions: Biological: pegfilgrastim; Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Arm V (Experimental): Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 4 courses. Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses. Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 3 hours on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.
  Interventions: Biological: pegfilgrastim; Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Arm VI (Experimental): Patients receive doxorubicin, cyclophosphamide, and pegfilgrastim as in arm V. Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 1 hour on day 1. Treatment repeats every 7 days for 12 courses.
  Interventions: Biological: pegfilgrastim; Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Biological: pegfilgrastim — Given IV
Drug: AC regimen — Given IV
Drug: cyclophosphamide — Given IV
Drug: doxorubicin hydrochloride — Given IV
Drug: paclitaxel — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and paclitaxel, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them after surgery may kill any remaining tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating resected breast cancer.

PURPOSE: This randomized phase III trial is comparing 2 different regimens of combination chemotherapy to see how well they work in treating patients who have undergone surgery for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival of patients with node-positive or high-risk node-negative breast cancer treated with 2 different schedules of adjuvant doxorubicin, cyclophosphamide, and paclitaxel.
* Compare the overall survival of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Correlate outcome with putative prognostic markers in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms (arms V and VI) (arms I-IV closed 11/10/10).

* Arm I: (closed 11/10/10) Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim subcutaneously (SC) on day 2 or filgrastim (G-CSF) SC on days 3-10. Treatment repeats every 14 days for 6 courses.

Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 3 hours on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.

* Arm II: (closed 11/10/10) Patients receive doxorubicin IV on day 1, oral cyclophosphamide on days 1-7, and G-CSF SC on days 2-7. Treatment repeats every 7 days for 15 courses.

Beginning 2 weeks after completion of cyclophosphamide, patients receive paclitaxel and pegfilgrastim as in arm I.

* Arm III: (closed 11/10/10) Patients receive doxorubicin, cyclophosphamide, and pegfilgrastim or G-CSF as in arm I.

Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 1 hour on day 1. Treatment repeats every 7 days for 12 courses.

* Arm IV: (closed 11/10/10) Patients receive doxorubicin, cyclophosphamide, and G-CSF as in arm II.

Beginning 2 weeks after completion of cyclophosphamide, patients receive paclitaxel as in arm III.

* Arm V: Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 4 courses. Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.

Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 3 hours on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.

* Arm VI: Patients receive doxorubicin, cyclophosphamide, and pegfilgrastim as in arm V.

Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 1 hour on day 1. Treatment repeats every 7 days for 12 courses.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

In all arms patients with HER2/neu-positive tumors also receive trastuzumab (Herceptin®) weekly or every 3 weeks beginning concurrently with paclitaxel OR 3 months after the last dose of paclitaxel and continuing for up to 52 weeks.

In all arms, patients with estrogen-receptor or progesterone-receptor positive tumors receive hormonal therapy beginning within 28 days of the completion of adjuvant chemotherapy or radiotherapy (if given).

After finishing study treatment patients are followed up every 6 months for 5 years and then once a year for up to 15 years.

PROJECTED ACCRUAL: A total of 3,250 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I-III invasive breast cancer

  * Operable disease
  * Stage I, II, IIIA, and IIIC (T1-3, N3a only)
  * No T4 tumors
* High-risk disease, defined by 1 of the following:

  * Tumor ≥ 2 cm in greatest diameter (includes both invasive and intraductal component)

    * Patients with nodal status of N0+ (i.e., no cluster of tumor cells in any node greater than 0.2 mm) are considered to be node negative and must have a primary tumor ≥ 2 cm in size or have a tumor ≥ 1 cm with high risk features
    * Patients who are node negative on the basis of a sentinel node procedure and fewer than 6 axillary nodes are removed are eligible OR at least 6 axillary or intramammary nodes must be negative
  * Tumor ≥ 1 cm in diameter and meeting 1 of the following criteria:

    * ER-negative and PgR-negative
    * ER-positive or PgR-positive with a Genomic Health Recurrence Score of ≥ 26
  * One or more axillary or intramammary nodes are involved by metastatic breast cancer

    * If one or more nodes is involved, a minimum of 6 axillary or intramammary nodes must have been examined histologically
    * Patients with N0(I+) disease will be considered node negative
* HER2/neu-positive tumors (3+ by immunohistochemical staining or amplified by fluorescence in-situ hybridization) allowed
* Bilateral synchronous breast cancer diagnosed within 1 month of each other allowed provided the higher TNM stage primary tumor meets the eligibility criteria
* Prior modified radical mastectomy OR local excision of all tumors with axillary lymph node dissection or sentinel node resection required

  * No more than 84 days since prior surgery for the primary tumor and/or axilla
  * Final resection margins for the primary tumor must be histologically negative for invasive cancer and ductal carcinoma in situ
  * Resection margins positive for lobular carcinoma in situ are allowed
* Hormone receptor status:

  * Estrogen receptor status known
  * Progesterone receptor status known

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* SGOT or SGPT no greater than 2 times ULN

Renal

* Creatinine no greater than ULN

Cardiovascular

* No congestive heart failure
* No active angina pectoris
* LVEF greater than or equal to the lower limit of normal* by MUGA or echocardiogram NOTE: Patients age 60 and over OR with a history of hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, in situ cervical carcinoma, or lobular carcinoma in situ of the breast

  * Prior invasive breast cancer or ductal carcinoma in situ allowed if disease-free for 5 years
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior cytotoxic chemotherapy for this breast cancer
* No prior chemotherapy with an anthracycline, anthracenedione, or taxane

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for this malignancy
* At least 2 weeks since prior radiotherapy for ductal carcinoma in situ

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3294 (Actual)
Dates: Start 2003-11; Primary Completion 2015-01 (Actual); Study Completion 2027-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: George Thomas Budd, MD, Study Chair — The Cleveland Clinic; Halle C Moore, MD, Study Director — The Cleveland Clinic
Locations (542):
- United States (539):
  - Regional Medical Center, Anniston, Alabama
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Sutter Solano Medical Center, Vallejo, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Kootenai Cancer Center - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - New Orleans Cancer Institute at Memorial Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Regional Cancer Center at Western Maryland Health System - Sacred Heart Campus, Cumberland, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Keesler Air Force Base Medical Center, Keesler Air Force Base, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Union State Bank Cancer Center at Nyack Hospital, Nyack, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital Cancer Treatment Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Cancer Care Associates at Troy and Dollie Smith Cancer Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - El Paso, El Paso, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Hematology-Oncology Associates of Fredericksburg, Incorporated, Fredericksburg, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (2):
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Budd GT, Barlow WE, Moore HC, Hobday TJ, Stewart JA, Isaacs C, Salim M, Cho JK, Rinn KJ, Albain KS, Chew HK, Burton GV, Moore TD, Srkalovic G, McGregor BA, Flaherty LE, Livingston RB, Lew DL, Gralow JR, Hortobagyi GN. SWOG S0221: a phase III trial comparing chemotherapy schedules in high-risk early-stage breast cancer. J Clin Oncol. 2015 Jan 1;33(1):58-64. doi: 10.1200/JCO.2014.56.3296. Epub 2014 Nov 24. PMID 25422488
- [Result] Sucheston LE, Zhao H, Yao S, Zirpoli G, Liu S, Barlow WE, Moore HC, Thomas Budd G, Hershman DL, Davis W, Ciupak GL, Stewart JA, Isaacs C, Hobday TJ, Salim M, Hortobagyi GN, Gralow JR, Livingston RB, Albain KS, Hayes DF, Ambrosone CB. Genetic predictors of taxane-induced neurotoxicity in a SWOG phase III intergroup adjuvant breast cancer treatment trial (S0221). Breast Cancer Res Treat. 2011 Dec;130(3):993-1002. doi: 10.1007/s10549-011-1671-3. Epub 2011 Jul 16. PMID 21766209
- [Result] Ambrosone CB, Sucheston LE, Zhao H, et al.: Variants in the BRCA1/Fanconi-anemia repair pathway and taxane-induced neuropathy in SWOG S0221. [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-2001, 2009.
- [Derived] Chen CS, Zirpoli G, Barlow WE, Budd GT, McKiver B, Pusztai L, Hortobagyi GN, Albain KS, Damaj MI, Godwin AK, Thompson A, Henry NL, Ambrosone CB, Stringer KA, Hertz DL. Vitamin D Insufficiency as a Risk Factor for Paclitaxel-Induced Peripheral Neuropathy in SWOG S0221. J Natl Compr Canc Netw. 2023 Nov;21(11):1172-1180.e3. doi: 10.6004/jnccn.2023.7062. PMID 37935109
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm V: (reopened in 12/2010) Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 4 courses. Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.
  Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 3 hours on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.
- Arm VI: (reopened in 12/2010) Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 4 courses. Patients receive doxorubicin IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2. Treatment repeats every 14 days for 6 courses.
  Beginning 2 weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 1 hour on day 1. Treatment repeats every 7 days for 12 courses.
Period: Overall Study
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Arm V | Arm VI
Started | 678 | 693 | 697 | 648 | 282 | 296
Completed | 478 | 490 | 526 | 481 | 203 | 244
Not Completed | 200 | 203 | 171 | 167 | 79 | 52
Not completed — Progression | 2 | 4 | 7 | 7 | 1 | 0
Not completed — Delinquent | 1 | 4 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 150 | 142 | 120 | 108 | 63 | 36
Not completed — Death | 4 | 1 | 5 | 3 | 0 | 1
Not completed — Other, not protocol specified | 17 | 15 | 14 | 19 | 6 | 7
Not completed — Withdrawal by Subject | 26 | 37 | 23 | 30 | 8 | 8
Not completed — Not reported | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only eligible and analyzable patients were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Arm V | ARM VI | Total
Number analyzed (Participants) | 664 | 683 | 681 | 639 | 277 | 294 | 3238
Age, Continuous [Median (Full Range); unit: years] | 50.5 [25 to 77] | 50.9 [23 to 79] | 51.8 [23 to 86] | 50.7 [21 to 76] | 52.7 [31 to 79] | 53.2 [23 to 76] | 52.7 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 658 | 679 | 676 | 636 | 275 | 291 | 3215
  Male | 6 | 4 | 5 | 3 | 2 | 3 | 23
Black Race [Count of Participants; unit: Participants] | 73 | 77 | 74 | 78 | 31 | 44 | 377
Menopausal status (females) [Count of Participants; unit: Participants] — Population: Only females of the total eligible and analyzable patients were included in menopausal status measurement.
  Participants
    number analyzed (Participants) | 658 | 679 | 676 | 636 | 275 | 291 | 3215
    Premenopausal | 326 | 325 | 308 | 299 | 124 | 123 | 1505
    Postmenopausal | 332 | 354 | 368 | 337 | 148 | 166 | 1705
    Unknown | 0 | 0 | 0 | 0 | 3 | 2 | 5
Nodal status [Count of Participants; unit: Participants]
  Negative | 161 | 153 | 159 | 146 | 105 | 109 | 833
  1-3 positive nodes | 260 | 266 | 276 | 245 | 103 | 98 | 1248
  >= 4 positive nodes | 241 | 264 | 243 | 244 | 68 | 87 | 1147
  unknown | 2 | 0 | 3 | 4 | 1 | 0 | 10
ER/PgR [Count of Participants; unit: Participants] — ER, estrogen receptor; PgR, progesterone receptor
  Participants
    Negative (both negative) | 212 | 226 | 232 | 206 | 99 | 108 | 1083
    Positive (either or both positive) | 450 | 456 | 446 | 430 | 178 | 185 | 2145
    Unknown | 2 | 1 | 3 | 3 | 0 | 1 | 10
HER2 [Count of Participants; unit: Participants] — HER2, human epidermal growth factor receptor 2.
  Participants
    Negative | 528 | 556 | 554 | 525 | 208 | 235 | 2606
    Positive | 125 | 123 | 118 | 109 | 69 | 57 | 601
    Unknown | 11 | 4 | 9 | 5 | 0 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Disease-free survival (DFS) defined as time from registration (randomization assignment) to first instance of disease recurrence (local, regional, or distant), new breast primary tumor, or death as a result of any cause. The results are entered as disease free survival at year 5.
Time Frame: every 6 months (annually for mammograms) for 5 years
Population: Only eligible and analyzable patients were included in this analysis. Two patients in Arm II and one patient in Arm IV with no follow-up were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Arm V | Arm VI
Number analyzed (Participants) | 664 | 681 | 681 | 638 | 277 | 294
percentage of participants | 83 [80 to 86] | 79 [76 to 82] | 81 [78 to 84] | 81 [78 to 84] | 84 [79 to 88] | 85 [80 to 89]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority or Other; p = 0.022, Log Rank; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.04 to 1.68]
Statistical Analysis 2: Comparison: Arm I vs Arm III; Test type: Superiority or Other; p = 0.072, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.98 to 1.59]
Statistical Analysis 3: Comparison: Arm I vs Arm IV; Test type: Superiority or Other; p = 0.38, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.87 to 1.44]
Statistical Analysis 4: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test type: Superiority or Other; p = 0.11, Log Rank
Statistical Analysis 5: Comparison: Arm V vs Arm VI; Test type: Superiority or Other; p = 0.733, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.61 to 1.41]

2. Primary Outcome: Overall Survival
Description: Overall survival defined as time from registration to death as result of any cause. Results were entered as overall survival rate at year 5.
Time Frame: Every 6 months for 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Arm V | Arm VI
Number analyzed (Participants) | 664 | 681 | 681 | 638 | 277 | 294
percentage of participants | 90 [87 to 92] | 87 [84 to 90] | 87 [84 to 89] | 87 [84 to 90] | 90 [86 to 93] | 91 [87 to 94]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority or Other; p = 0.013, Log Rank; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [1.08 to 1.93]
Statistical Analysis 2: Comparison: Arm I vs Arm III; Test type: Superiority or Other; p = 0.011, Log Rank; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [1.09 to 1.95]
Statistical Analysis 3: Comparison: Arm I vs Arm IV; Test type: Superiority or Other; p = 0.17, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.91 to 1.68]
Statistical Analysis 4: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test type: Superiority or Other; p = 0.040, Log Rank
Statistical Analysis 5: Comparison: Arm V vs Arm VI; Test type: Superiority or Other; p = 0.724, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.54 to 1.53]

3. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 3.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Toxicity assessment was evaluated every 4 weeks while on protocol therapy.
Population: Limited to patients who started treatment, who did not have a major deviation in the treatment protocol, and whose toxicity profile has been completed.
Measure: Number; unit: Participants
Arm/Group | ARM I | ARM II | ARM III | ARM IV | ARM V | ARM VI
Number analyzed (Participants) | 654 | 663 | 674 | 624 | 275 | 291
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 7 | 4 | 3 | 4 | 3 | 1
  AST, SGOT | 5 | 3 | 2 | 2 | 4 | 1
  Acidosis (metabolic or respiratory) | 1 | 0 | 0 | 0 | 0 | 0
  Adult respiratory distress syndrome (ARDS) | 1 | 0 | 2 | 0 | 0 | 1
  Albumin, serum-low (hypoalbuminemia) | 1 | 2 | 0 | 0 | 0 | 0
  Alkaline phosphatase | 0 | 0 | 0 | 1 | 0 | 0
  Allergic reaction/hypersensitivity | 8 | 12 | 6 | 3 | 5 | 5
  Anorexia | 6 | 5 | 8 | 4 | 0 | 2
  Apnea | 0 | 0 | 1 | 0 | 0 | 0
  Arthritis (non-septic) | 0 | 0 | 0 | 0 | 0 | 1
  Ataxia (incoordination) | 2 | 0 | 1 | 0 | 0 | 0
  Bilirubin (hyperbilirubinemia) | 3 | 0 | 2 | 0 | 0 | 0
  Bladder spasms | 0 | 2 | 0 | 0 | 0 | 0
  Blood/Bone Marrow-Other | 1 | 2 | 2 | 0 | 0 | 0
  Bronchospasm, wheezing | 0 | 1 | 0 | 0 | 1 | 0
  CNS cerebrovascular ischemia | 0 | 0 | 1 | 1 | 0 | 0
  Calcium, serum-high (hypercalcemia) | 0 | 0 | 0 | 1 | 0 | 0
  Calcium, serum-low (hypocalcemia) | 2 | 1 | 1 | 0 | 1 | 1
  Cardiac General-Other | 2 | 1 | 1 | 0 | 0 | 0
  Cardiac troponin I (cTnI) | 0 | 0 | 1 | 1 | 0 | 0
  Cardiac troponin T (cTnT) | 3 | 0 | 2 | 0 | 0 | 0
  Cardiac-ischemia/infarction | 3 | 0 | 1 | 0 | 1 | 0
  Cardiopulmonary arrest, cause unknown (non-fatal) | 0 | 0 | 1 | 0 | 0 | 0
  Cataract | 0 | 1 | 0 | 0 | 0 | 0
  Cholecystitis | 1 | 0 | 0 | 0 | 0 | 0
  Colitis | 1 | 0 | 2 | 1 | 1 | 0
  Colitis, infectious (e.g., Clostridium difficile) | 0 | 0 | 1 | 2 | 0 | 0
  Conduction abnormality - Asystole | 0 | 0 | 1 | 0 | 0 | 0
  Confusion | 1 | 1 | 0 | 0 | 0 | 1
  Constipation | 3 | 3 | 3 | 3 | 1 | 0
  Constitutional Symptoms-Other | 1 | 1 | 0 | 0 | 0 | 0
  Cough | 3 | 5 | 4 | 0 | 1 | 1
  Creatinine | 1 | 0 | 0 | 0 | 0 | 0
  Cystitis | 0 | 3 | 0 | 0 | 0 | 0
  Cytokine release syndrome/acute infusion reaction | 0 | 0 | 0 | 2 | 1 | 0
  DIC (disseminated intravascular coagulation) | 1 | 0 | 0 | 0 | 0 | 0
  Death - Multi-organ failure | 1 | 0 | 1 | 0 | 0 | 0
  Death not associated with CTCAE term - Death NOS | 0 | 0 | 0 | 1 | 0 | 1
  Dehydration | 8 | 7 | 12 | 3 | 4 | 4
  Dermatology/Skin-Other | 0 | 3 | 0 | 1 | 1 | 0
  Diarrhea | 27 | 18 | 24 | 23 | 8 | 6
  Distention/bloating, abdominal | 0 | 0 | 1 | 1 | 0 | 0
  Dizziness | 5 | 2 | 2 | 5 | 0 | 2
  Dysphagia (difficulty swallowing) | 2 | 0 | 1 | 3 | 0 | 0
  Dyspnea (shortness of breath) | 21 | 18 | 25 | 16 | 2 | 4
  Edema: head and neck | 0 | 1 | 0 | 0 | 0 | 0
  Edema: limb | 0 | 2 | 2 | 3 | 1 | 1
  Encephalopathy | 1 | 0 | 0 | 0 | 0 | 0
  Endocrine-Other | 0 | 0 | 1 | 0 | 0 | 0
  Esophagitis | 5 | 4 | 0 | 3 | 0 | 0
  Extrapyramidal/involuntary movement/restlessness | 0 | 0 | 0 | 1 | 0 | 0
  Extremity-upper (function) | 0 | 0 | 1 | 0 | 0 | 0
  Eyelid dysfunction | 0 | 0 | 0 | 0 | 1 | 0
  FEV(1) | 0 | 0 | 1 | 0 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 77 | 59 | 87 | 65 | 20 | 14
  Febrile neutropenia | 49 | 9 | 38 | 20 | 16 | 14
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 2 | 3 | 3 | 1 | 1 | 1
  Fistula, GI - Oral cavity | 0 | 0 | 0 | 1 | 0 | 0
  Flu-like syndrome | 0 | 1 | 1 | 1 | 0 | 0
  Fracture | 0 | 2 | 0 | 0 | 0 | 2
  GGT (gamma-glutamyl transpeptidase) | 2 | 0 | 0 | 1 | 0 | 0
  Gastritis (including bile reflux gastritis) | 0 | 0 | 0 | 1 | 0 | 0
  Gastrointestinal-Other | 1 | 0 | 0 | 3 | 0 | 0
  Glucose, serum-high (hyperglycemia) | 13 | 17 | 9 | 13 | 6 | 5
  Glucose, serum-low (hypoglycemia) | 4 | 2 | 0 | 1 | 0 | 0
  Hair loss/Alopecia (scalp or body) | 3 | 0 | 0 | 0 | 0 | 0
  Heartburn/dyspepsia | 1 | 0 | 3 | 5 | 1 | 1
  Hemoglobin | 87 | 48 | 101 | 47 | 21 | 19
  Hemorrhage, GI - Lower GI NOS | 0 | 1 | 0 | 1 | 1 | 0
  Hemorrhage, GI - Oral cavity | 0 | 0 | 0 | 1 | 0 | 0
  Hemorrhage, GI - Rectum | 1 | 0 | 0 | 0 | 1 | 0
  Hemorrhage, GI - Upper GI NOS | 1 | 0 | 0 | 0 | 0 | 0
  Hemorrhage, GU - Urinary NOS | 0 | 0 | 0 | 1 | 0 | 0
  Hemorrhage, GU - Vagina | 0 | 0 | 1 | 0 | 0 | 0
  Hemorrhage, pulmonary/upper respiratory - Nose | 0 | 0 | 0 | 1 | 0 | 1
  Hemorrhage/Bleeding-Other | 1 | 0 | 0 | 1 | 0 | 0
  Hemorrhoids | 1 | 3 | 1 | 0 | 0 | 1
  Hot flashes/flushes | 0 | 2 | 1 | 0 | 1 | 1
  Hypertension | 2 | 1 | 1 | 1 | 2 | 2
  Hypotension | 4 | 1 | 4 | 3 | 0 | 3
  Hypoxia | 2 | 3 | 3 | 2 | 3 | 1
  INR (of prothrombin time) | 2 | 5 | 1 | 3 | 1 | 2
  Ileus, GI (functional obstruction of bowel) | 0 | 0 | 1 | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Abdomen NOS | 0 | 1 | 0 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Bladder | 0 | 1 | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 2 | 1 | 2 | 0 | 2 | 3
  Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel | 0 | 1 | 0 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 0 | 0 | 0 | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Eye NOS | 0 | 0 | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 4 | 2 | 2 | 4 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lymphatic | 0 | 0 | 2 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Meninges | 0 | 0 | 0 | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Middle ear | 0 | 0 | 1 | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Mucosa | 1 | 1 | 0 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 0 | 0 | 1 | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Paranasal | 0 | 0 | 0 | 2 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Pharynx | 0 | 0 | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 3 | 1 | 2 | 3 | 1 | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Soft tissue | 0 | 0 | 0 | 0 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1 | 2 | 0 | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 0 | 0 | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Wound | 0 | 2 | 3 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Bil. tree | 0 | 0 | 0 | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Bladder | 0 | 1 | 1 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2 | 0 | 0 | 2 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus | 0 | 2 | 0 | 2 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Catheter | 0 | 2 | 2 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Colon | 0 | 0 | 1 | 1 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Dental | 0 | 1 | 0 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Esophagus | 0 | 0 | 0 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Kidney | 1 | 1 | 0 | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 7 | 5 | 10 | 5 | 2 | 4
  Inf w/normal ANC or Gr 1-2 neutrophils - Meninges | 2 | 0 | 0 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Muscle | 0 | 0 | 0 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Neck NOS | 0 | 1 | 0 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Oral cav | 1 | 0 | 0 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Sinus | 2 | 2 | 2 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 7 | 6 | 8 | 11 | 4 | 4
  Inf w/normal ANC or Gr 1-2 neutrophils - Soft tiss | 1 | 0 | 1 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 5 | 3 | 0 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Ungual | 0 | 1 | 1 | 2 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Up airway | 0 | 1 | 2 | 2 | 1 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Vagina | 0 | 1 | 0 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Vulva | 1 | 0 | 0 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Wound | 0 | 1 | 0 | 2 | 1 | 3
  Inf w/normal ANC or Gr 1-2 neutrophils - perioral | 0 | 0 | 1 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils -Nerve-cran | 0 | 0 | 1 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils-Foreign bod | 0 | 1 | 0 | 0 | 0 | 1
  Infection with normal ANC or Grade 1 or 2 neutroph | 1 | 0 | 1 | 1 | 0 | 0
  Infection with unknown ANC - Appendix | 1 | 0 | 0 | 0 | 0 | 0
  Infection with unknown ANC - Blood | 0 | 0 | 0 | 0 | 0 | 1
  Infection with unknown ANC - Catheter-related | 0 | 1 | 0 | 0 | 0 | 0
  Infection with unknown ANC - Foreign body (e.g., g | 0 | 0 | 0 | 0 | 0 | 1
  Infection with unknown ANC - Kidney | 0 | 0 | 0 | 1 | 0 | 0
  Infection with unknown ANC - Lung (pneumonia) | 0 | 1 | 0 | 0 | 1 | 0
  Infection with unknown ANC - Skin (cellulitis) | 1 | 0 | 0 | 0 | 0 | 1
  Infection with unknown ANC - Wound | 0 | 0 | 0 | 0 | 1 | 0
  Infection-Other | 4 | 3 | 5 | 0 | 2 | 1
  Injection site reaction/extravasation changes | 1 | 0 | 1 | 0 | 0 | 0
  Insomnia | 1 | 1 | 0 | 6 | 1 | 1
  Intra-operative injury - Peripheral sensory NOS | 0 | 0 | 0 | 0 | 0 | 2
  Intra-operative injury - Spinal cord | 0 | 0 | 0 | 1 | 0 | 0
  Irregular menses (change from baseline) | 1 | 1 | 0 | 0 | 0 | 0
  Joint-function | 0 | 1 | 0 | 0 | 0 | 0
  Left ventricular diastolic dysfunction | 3 | 0 | 3 | 0 | 0 | 0
  Left ventricular systolic dysfunction | 7 | 2 | 8 | 2 | 1 | 1
  Leukocytes (total WBC) | 128 | 98 | 157 | 128 | 38 | 34
  Liver dysfunction/failure (clinical) | 1 | 0 | 1 | 0 | 0 | 0
  Lymphopenia | 24 | 31 | 26 | 32 | 15 | 18
  Magnesium, serum-low (hypomagnesemia) | 0 | 0 | 1 | 0 | 0 | 0
  Metabolic/Laboratory-Other | 1 | 0 | 0 | 0 | 0 | 0
  Mood alteration - agitation | 1 | 0 | 0 | 0 | 0 | 0
  Mood alteration - anxiety | 1 | 2 | 1 | 0 | 0 | 0
  Mood alteration - depression | 1 | 6 | 4 | 4 | 1 | 2
  Mucositis/stomatitis (clinical exam) - Anus | 0 | 1 | 0 | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Esophagus | 1 | 0 | 0 | 2 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 17 | 56 | 23 | 57 | 4 | 3
  Mucositis/stomatitis (clinical exam) - Pharynx | 2 | 5 | 3 | 1 | 0 | 0
  Mucositis/stomatitis (functional/symp) - Anus | 0 | 1 | 0 | 0 | 0 | 0
  Mucositis/stomatitis (functional/symp) - Esophagus | 2 | 3 | 2 | 5 | 1 | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 11 | 38 | 28 | 40 | 1 | 6
  Mucositis/stomatitis (functional/symp) - Pharynx | 4 | 4 | 5 | 4 | 0 | 1
  Mucositis/stomatitis (functional/symp) - Rectum | 1 | 0 | 0 | 0 | 0 | 0
  Muscle weakness, not d/t neuropathy - Extrem-lower | 0 | 0 | 0 | 0 | 2 | 1
  Muscle weakness, not d/t neuropathy - body/general | 0 | 1 | 1 | 2 | 1 | 1
  Musculoskeletal/Soft Tissue-Other | 1 | 0 | 0 | 0 | 0 | 0
  Myelodysplasia | 0 | 1 | 1 | 0 | 0 | 0
  Myocarditis | 0 | 0 | 1 | 0 | 0 | 1
  Nail changes | 4 | 12 | 5 | 9 | 1 | 1
  Nasal cavity/paranasal sinus reactions | 1 | 0 | 0 | 0 | 0 | 0
  Nausea | 50 | 40 | 53 | 33 | 9 | 9
  Neurology-Other | 0 | 1 | 0 | 0 | 0 | 0
  Neuropathy: CN V Motor-jaw muscles; Sensory-facial | 1 | 0 | 1 | 1 | 0 | 0
  Neuropathy: CN VII Motor-face; Sensory-taste | 1 | 0 | 0 | 0 | 0 | 1
  Neuropathy: cranial - CN VIII Hearing and balance | 0 | 0 | 0 | 1 | 0 | 0
  Neuropathy: cranial - CN XII Motor-tongue | 1 | 0 | 0 | 0 | 0 | 0
  Neuropathy: motor | 10 | 13 | 8 | 6 | 5 | 8
  Neuropathy: sensory | 107 | 101 | 76 | 56 | 45 | 25
  Neutrophils/granulocytes (ANC/AGC) | 174 | 156 | 218 | 201 | 57 | 65
  Obesity | 0 | 0 | 0 | 0 | 1 | 3
  Obstruction, GI - Small bowel NOS | 0 | 1 | 0 | 0 | 0 | 0
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 0 | 0 | 1 | 0 | 0 | 0
  PTT (Partial thromboplastin time) | 0 | 1 | 0 | 0 | 0 | 0
  Pain - Abdomen NOS | 2 | 3 | 5 | 0 | 5 | 2
  Pain - Anus | 1 | 1 | 0 | 0 | 0 | 0
  Pain - Back | 0 | 5 | 1 | 3 | 2 | 2
  Pain - Bone | 10 | 36 | 15 | 9 | 15 | 1
  Pain - Breast | 0 | 0 | 0 | 0 | 0 | 2
  Pain - Cardiac/heart | 1 | 0 | 0 | 1 | 1 | 0
  Pain - Chest wall | 1 | 0 | 0 | 0 | 1 | 0
  Pain - Chest/thorax NOS | 0 | 1 | 0 | 3 | 0 | 0
  Pain - Dental/teeth/peridontal | 0 | 1 | 0 | 0 | 0 | 1
  Pain - Esophagus | 0 | 0 | 0 | 1 | 0 | 0
  Pain - Extremity-limb | 4 | 9 | 0 | 3 | 4 | 1
  Pain - Head/headache | 5 | 8 | 10 | 10 | 1 | 0
  Pain - Joint | 39 | 40 | 21 | 12 | 11 | 5
  Pain - Kidney | 0 | 0 | 0 | 2 | 0 | 0
  Pain - Middle ear | 0 | 1 | 0 | 1 | 0 | 0
  Pain - Muscle | 42 | 48 | 21 | 11 | 10 | 5
  Pain - Neck | 0 | 1 | 0 | 0 | 0 | 1
  Pain - Neuralgia/peripheral nerve | 1 | 3 | 2 | 3 | 1 | 0
  Pain - Pain NOS | 3 | 0 | 0 | 1 | 0 | 1
  Pain - Pelvis | 0 | 1 | 0 | 0 | 0 | 0
  Pain - Rectum | 2 | 1 | 0 | 2 | 0 | 0
  Pain - Skin | 0 | 1 | 0 | 0 | 0 | 0
  Pain - Stomach | 0 | 0 | 0 | 1 | 0 | 0
  Pain - Uterus | 0 | 0 | 0 | 0 | 1 | 0
  Pain-Other | 3 | 5 | 2 | 1 | 4 | 0
  Pericardial effusion (non-malignant) | 0 | 0 | 0 | 0 | 0 | 2
  Phosphate, serum-low (hypophosphatemia) | 0 | 3 | 0 | 2 | 0 | 0
  Platelets | 24 | 21 | 20 | 22 | 6 | 2
  Pleural effusion (non-malignant) | 0 | 1 | 1 | 0 | 0 | 1
  Pneumonitis/pulmonary infiltrates | 8 | 7 | 11 | 5 | 3 | 1
  Potassium, serum-high (hyperkalemia) | 1 | 1 | 0 | 1 | 0 | 0
  Potassium, serum-low (hypokalemia) | 18 | 12 | 18 | 7 | 8 | 8
  Prolapse of stoma, GI | 2 | 3 | 2 | 4 | 0 | 0
  Proteinuria | 0 | 1 | 0 | 0 | 0 | 0
  Pruritus/itching | 2 | 3 | 0 | 1 | 2 | 1
  Psychosis (hallucinations/delusions) | 0 | 0 | 1 | 0 | 0 | 0
  Pulmonary/Upper Respiratory-Other | 1 | 2 | 1 | 0 | 1 | 1
  Rash/desquamation | 4 | 5 | 1 | 4 | 1 | 1
  Rash: acne/acneiform | 0 | 0 | 1 | 0 | 0 | 0
  Rash: hand-foot skin reaction | 19 | 95 | 16 | 94 | 3 | 4
  Restrictive cardiomyopathy | 0 | 0 | 1 | 1 | 0 | 0
  Right ventricular dysfunction (cor pulmonale) | 0 | 1 | 0 | 0 | 0 | 0
  Rigors/chills | 1 | 0 | 0 | 0 | 0 | 0
  SVT and nodal arrhythmia - Atrial fibrillation | 1 | 1 | 5 | 1 | 0 | 0
  SVT and nodal arrhythmia - SVT tachycardia | 0 | 1 | 0 | 0 | 0 | 0
  SVT and nodal arrhythmia - Sinus tachycardia | 0 | 1 | 1 | 0 | 0 | 0
  Salivary gland changes/saliva | 0 | 1 | 0 | 0 | 0 | 0
  Secondary Malignancy-poss rel to cancer Tx | 2 | 2 | 4 | 3 | 1 | 0
  Seizure | 0 | 1 | 1 | 1 | 0 | 1
  Seroma | 0 | 0 | 2 | 0 | 0 | 0
  Sodium, serum-high (hypernatremia) | 1 | 0 | 0 | 0 | 0 | 0
  Sodium, serum-low (hyponatremia) | 7 | 4 | 5 | 4 | 1 | 3
  Somnolence/depressed level of consciousness | 2 | 1 | 0 | 1 | 0 | 2
  Sudden death | 2 | 0 | 0 | 0 | 0 | 0
  Syncope (fainting) | 5 | 5 | 7 | 5 | 5 | 7
  Syndromes-Other | 0 | 2 | 1 | 0 | 0 | 0
  Taste alteration (dysgeusia) | 1 | 0 | 2 | 0 | 0 | 0
  Thrombosis/embolism (vascular access-related) | 9 | 18 | 10 | 6 | 1 | 4
  Thrombosis/thrombus/embolism | 10 | 7 | 9 | 8 | 3 | 4
  Ulcer, GI - Esophagus | 1 | 0 | 0 | 0 | 0 | 0
  Ulcer, GI - Rectum | 0 | 0 | 0 | 0 | 1 | 0
  Uric acid, serum-high (hyperuricemia) | 1 | 0 | 0 | 0 | 0 | 0
  Urticaria (hives, welts, wheals) | 1 | 0 | 0 | 0 | 0 | 1
  Vaginitis (not due to infection) | 0 | 0 | 0 | 1 | 0 | 0
  Valvular heart disease | 1 | 0 | 0 | 0 | 0 | 0
  Vasovagal episode | 0 | 0 | 1 | 0 | 0 | 0
  Ventricular arrhythmia - PVCs | 1 | 0 | 0 | 0 | 0 | 0
  Ventricular arrhythmia - Ventricular tachycardia | 1 | 1 | 1 | 0 | 0 | 0
  Viral hepatitis | 1 | 0 | 0 | 0 | 0 | 1
  Vision-blurred vision | 1 | 0 | 1 | 2 | 0 | 0
  Voice changes/dysarthria | 0 | 0 | 0 | 0 | 0 | 1
  Vomiting | 31 | 29 | 38 | 17 | 8 | 6
  Watery eye (epiphora, tearing) | 0 | 2 | 0 | 0 | 0 | 0
  Weight loss | 2 | 2 | 1 | 1 | 0 | 2
  Wound complication, non-infectious | 0 | 1 | 1 | 0 | 1 | 0

4. Secondary Outcome: Disease-free Survival Comparison Between 2 Treatments in HR-positive, HER-2 Negative Group
Description: as for outcome 1
Time Frame: Biomarkers were measured by gene expression analysis before study entry. DFS were measured every 6 months for 5 years
Population: Patients with HR-positive, HER-2 negative at baseline in each arm were included in this analysis. Arm V and Arm VI were reopened under a new revised protocol and the data were not mature. And the results for Arm V and Arm VI will be reported in a subsequent publication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 375 | 370 | 373 | 362
percentage of participants | 82 [78 to 86] | 82 [77 to 86] | 86 [82 to 89] | 85 [80 to 88]
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Overall treatment differences; Test type: Superiority or Other; p = 0.67, Log Rank
Statistical Analysis 2: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of interaction of two treatments: AC and paclitaxel; Test type: Superiority or Other; p = 0.42, Log Rank

5. Secondary Outcome: Overall Survival Comparison Between 2 Treatments in HR-positive, HER-2 Negative Group
Description: as for outcome 2
Time Frame: Biomarkers were measured by gene expression analysis before study entry. OS was measured every 6 months for 5 years
Population: Patients with HR-positive, HER-negative at baseline in each arm were included in this analysis. Arm V and Arm VI were reopened under a new revised protocol and the data were not mature. And the results for Arm V and Arm VI will be reported in a subsequent publication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 375 | 370 | 373 | 362
percentage of participants | 91 [87 to 93] | 92 [89 to 95] | 91 [87 to 94] | 90 [86 to 93]
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of overall treatment differences; Test type: Superiority or Other; p = 0.90, Log Rank
Statistical Analysis 2: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of interaction of two treatments: AC and paclitaxel; Test type: Superiority or Other; p = 0.52, Log Rank

6. Secondary Outcome: Disease-free Survival Comparison Between 2 Treatments in HR-negative, HER-2 Negative Group
Description: as for outcome 1
Time Frame: Biomarkers were measured by gene expression analysis before study entry. DFS was measured every 6 months for 5 years
Population: Patients with HR-negative, HER-2 negative at baseline in each arm were included in this analysis. Arm V and Arm VI were reopened under a new revised protocol and the data were not mature. And the results for Arm V and Arm VI will be reported in a subsequent publication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 153 | 185 | 180 | 162
percentage of participants | 83 [75 to 88] | 71 [63 to 77] | 72 [64 to 78] | 75 [68 to 81]
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of overall treatment differences; Test type: Superiority or Other; p = 0.076, Log Rank
Statistical Analysis 2: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of interaction of two treatments: AC and paclitaxel; Test type: Superiority or Other; p = 0.018, Log Rank

7. Secondary Outcome: Overall Survival Comparison Between 2 Treatments in HR-negative, HER-2 Negative Group
Description: as for outcome 2
Time Frame: Biomarkers were measured by gene expression analysis before study entry. OS was measured every 6 months for 5 years
Population: Patients with HR-negative, HER2-negative at baseline in each arm were included in this analysis. Arm V and Arm VI were reopened under a new revised protocol and the data were not mature. And the results for Arm V and Arm VI will be reported in a subsequent publication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 153 | 185 | 180 | 162
percentage of participants | 85 [78 to 90] | 76 [69 to 82] | 78 [71 to 84] | 82 [75 to 87]
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of overall treatment differences; Test type: Superiority or Other; p = 0.062, Log Rank
Statistical Analysis 2: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of interaction of two treatments: AC and paclitaxel; Test type: Superiority or Other; p = 0.010, Log Rank

8. Secondary Outcome: Disease-free Survival Comparison Between 2 Treatments in HER2-positive Group
Description: as for outcome 1
Time Frame: Biomarkers were measured by gene expression analysis before study entry. DFS was measured every 6 months for 5 years
Population: Patients with HER2-positive at baseline in each arm were included in this analysis. One patient in Arm II with no follow-up was excluded. Arm V and Arm VI were reopened under a new revised protocol and the data were not mature. And the results for Arm V and Arm VI will be reported in a subsequent publication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 125 | 122 | 118 | 109
percentage of participants | 85 [77 to 90] | 83 [74 to 89] | 82 [74 to 88] | 80 [71 to 87]
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of overall treatment differences; Test type: Superiority or Other; p = 0.69, Log Rank
Statistical Analysis 2: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of interaction two treatments: AC and paclitaxel; Test type: Superiority or Other; p = 0.66, Log Rank

9. Secondary Outcome: Overall Survival Comparison Between 2 Treatments in HER-2 Positive Group.
Description: as for outcome 2
Time Frame: Biomarkers were measured by gene expression analysis before study entry. OS was measured every 6 months for 5 years
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 125 | 122 | 118 | 109
percentage of participants | 94 [88 to 97] | 89 [81 to 94] | 89 [82 to 94] | 88 [80 to 93]
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of overall treatment differences; Test type: Superiority or Other; p = 0.40, Log Rank
Statistical Analysis 2: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Test of interaction of two treatments: AC and paclitaxel; Test type: Superiority or Other; p = 0.28, Log Rank

ADVERSE EVENTS:
Time Frame: Toxicity assessment was evaluated every 4 weeks while on protocol therapy.
Arm/Group | ARM I | ARM II | ARM III | ARM IV | ARM V | ARM VI
Serious Adverse Events (participants affected / at risk) | 10/654 | 8/663 | 17/674 | 9/624 | 5/275 | 8/291
Other Adverse Events (participants affected / at risk) | 381/654 | 412/663 | 389/674 | 391/624 | 131/275 | 126/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM I (N=654) | ARM II (N=663) | ARM III (N=674) | ARM IV (N=624) | ARM V (N=275) | ARM VI (N=291)
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Cardiac-ischemia/infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conduction abnormality - Asystole (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular arrhythmia - PVCs (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constitutional Symptoms-Other (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Death - Multi-organ failure (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Death not associated with CTCAE term - Death NOS (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Soft tiss (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
AST, SGOT (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac troponin I (cTnI) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 0 | 1 | 0 | 3 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Secondary Malignancy-poss rel to cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 4 | 3 | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 2 | 2 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARM I (N=654) | ARM II (N=663) | ARM III (N=674) | ARM IV (N=624) | ARM V (N=275) | ARM VI (N=291)
Febrile neutropenia (Blood and lymphatic system disorders) | 49 | 9 | 38 | 20 | 15 | 12
Hemoglobin (Blood and lymphatic system disorders) | 87 | 48 | 101 | 47 | 21 | 19
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 17 | 56 | 23 | 57 | 4 | 3
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 11 | 38 | 28 | 40 | 1 | 6
Nausea (Gastrointestinal disorders) | 50 | 40 | 53 | 33 | 9 | 9
Vomiting (Gastrointestinal disorders) | 31 | 29 | 38 | 17 | 8 | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 77 | 59 | 87 | 65 | 20 | 14
Leukocytes (total WBC) (Investigations) | 128 | 98 | 157 | 128 | 38 | 34
Lymphopenia (Investigations) | 24 | 31 | 26 | 32 | 15 | 18
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 174 | 156 | 217 | 201 | 54 | 65
Pain - Bone (Musculoskeletal and connective tissue disorders) | 10 | 36 | 15 | 9 | 15 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 39 | 40 | 21 | 12 | 11 | 5
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 42 | 48 | 21 | 11 | 10 | 5
Neuropathy: sensory (Nervous system disorders) | 107 | 101 | 76 | 56 | 45 | 25
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 19 | 95 | 16 | 94 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less